CLINICAL TRIAL: NCT07128199
Title: A Randomized, Placebo-Controlled, Double-Blind, Multi-Center Phase 3 Study of Zipalertinib Plus Adjuvant Chemotherapy Versus Placebo Plus Adjuvant Chemotherapy in Stage IB-IIIA NSCLC Patients With Uncommon EGFR Mutations Following Complete Tumor Resection (REZILIENT4)
Brief Title: A Study to Assess the Efficacy and Safety of Zipalertinib Versus Placebo for Adjuvant Treatment in Participants With Stage IB-IIIA NSCLC With Uncommon EGFR Mutations, Following Complete Tumor Resection
Acronym: REZILIENT4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAS6417-302; 2025-521775-31-00 (Other: EU Trial Number)
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: NSCLC, Stage IB-IIIA; Lung Cancer; Adjuvant; Post-surgical; EGFR; Exon 20; Early Stage Lung Cancer; Uncommon EGFR Mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cisplatin; Carboplatin; Pemetrexed; zipalertinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zipalertinib (Experimental): Participants will receive adjuvant platinum-based chemotherapy consisting of cisplatin 75 milligrams per square meter (mg/m^2) or carboplatin (area under concentration [AUC] 5 milligrams per milliliter per minute mg/mL/min) plus pemetrexed 500 mg/m^2, administered via intravenous (IV) infusion, on 21-day cycle, in combination with zipalertinib 100 mg, orally, twice daily (BID).
  After completion of chemotherapy, participants will continue on zipalertinib monotherapy 100 mg, orally, BID on 21-day cycle, until the participant meets any of the treatment discontinuation criteria.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: TAS6417
- Placebo (Placebo Comparator): Participants will receive adjuvant platinum-based chemotherapy consisting of cisplatin 75 mg/m^2 or carboplatin AUC 5 mg/mL/min plus pemetrexed 500 mg/m^2, administered via IV infusion, on 21-day cycle, in combination with zipalertinib matching-placebo 100 mg, orally, BID.
  After completion of chemotherapy, participants will continue on zipalertinib matching-placebo monotherapy 100mg, orally, BID on 21-day cycle, until the participant meets any of the treatment discontinuation criteria.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Zipalertinib Matching-placebo

INTERVENTIONS:
Drug: Cisplatin — IV infusion.
Drug: Carboplatin — IV infusion.
Drug: Pemetrexed — IV infusion.
Drug: TAS6417 — Oral tablets.
  Other Names: Zipalertinib; CLN-081
  Arms: Zipalertinib
Drug: Zipalertinib Matching-placebo — Oral tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of zipalertinib combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in participants with early stage (stage IB-IIIA) resected non-small cell lung cancer (NSCLC) harboring uncommon epidermal growth factor receptor mutation (EGFRmt).

DETAILED DESCRIPTION:
This study will evaluate zipalertinib, a novel EGFR tyrosine kinase inhibitor (TKI) in combination with standard platinum-based adjuvant chemotherapy versus placebo in combination with chemotherapy in participants with resected stage IB-IIIA NSCLC harboring uncommon EGFRmt.

Approximately 360 participants will be randomized 1:1 to:

Arm A: Platinum-based chemotherapy (cisplatin or carboplatin plus pemetrexed) in combination with zipalertinib 100 milligrams (mg) twice daily (BID), followed by zipalertinib 100 mg BID alone OR

Arm B: Platinum-based chemotherapy (cisplatin or carboplatin plus pemetrexed) in combination with placebo BID, followed by placebo BID alone.

The duration of 1 treatment cycle will be 21 days. An independent data monitoring committee (IDMC) will be established to monitor interim safety data.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of primary NSCLC on predominantly non-squamous histology.
2. Documented EGFRmt status as determined by local testing performed at a clinical laboratory improvement amendment (CLIA) certified (United States [US]) or accredited (outside of the US) local laboratory, defined as either one of the following EGFRmt:

   1. exon20 insertion mutations (ex20ins) or
   2. other uncommon, non-ex20ins EGFRmt (eg, G719X, L861Q, or S768I)
3. Magnetic resonance imaging (MRI) or computed tomography (CT) scan of the brain done prior to surgery. Participants in whom this was not done prior to surgery may still be enrolled if appropriate imaging (i.e., MRI or CT of the brain) is performed prior to randomization.
4. Complete surgical resection of the primary NSCLC is mandatory. All gross disease must have been removed at the end of surgery. All surgical margins of resection must be negative for tumor. Resection may be accomplished by open thoracotomy or video associated thoracic surgery (VATS) techniques.
5. Classified post-operatively as either Stage IB, IIA, IIB, or IIIA according to the tumor nodes metastasis (TNM) staging system for lung cancer (American Joint Committee on Cancer [AJCC] 9th edition).
6. Complete recovery from surgery at the time of randomization.
7. Eastern cooperative oncology group performance status (ECOG PS) of 0 or 1.
8. Archival tumor tissue available for submission, with minimum quantity sufficient to evaluate EGFRmt status and, where possible, other biomarkers.

Exclusion Criteria:

1. Is currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Treatment with any of the following within the time frame specified:

   1. Zipalertinib (TAS6417/CLN-081) or any other EGFR inhibitor at any time.
   2. Pre-operative or post-operative or planned radiation therapy for the current lung cancer.
   3. Any prior systemic anticancer therapy (e.g., neoadjuvant chemotherapy), including investigational therapy, for treatment of NSCLC.
   4. Major surgery (including primary tumor surgery, excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
   5. All prescribed medication, over-the-counter medication, vitamin preparations and other food supplements, or herbal medications that are strong or moderate cytochrome p450 (CYP) 3A4 inducers or inhibitors within 7 days prior to first dose.
   6. Treatment with an investigational drug within five half-lives of the compound or any of its related material, if known.
3. Has received only segmentectomies or wedge resections.
4. Past medical history of interstitial lung disease (ILD)/pneumonitis, drug-induced ILD/pneumonitis or any evidence of clinically active ILD/pneumonitis.
5. Impaired cardiac function or clinically significant cardiac disease.
6. Unable to swallow tablets or has any disease or condition that may significantly affect gastrointestinal (GI) absorption of zipalertinib (such as inflammatory bowel disease, malabsorption syndrome, or prior significant bowel resection).
7. Participants with a history of any other cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, other cancers curatively treated with no evidence of disease for >5 years following the end of treatment and which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
8. Known history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) that is unstable or not controlled with treatment. Screening not required.
9. Active bleeding disorders.
10. Known:

    a. Hypersensitivity: i. To the ingredients in zipalertinib/placebo or any drugs similar in structure or class. ii. To platinum-containing drugs (i.e., cisplatin, carboplatin), pemetrexed, or any known excipients of these drugs. b. Contraindications to platinum-containing drugs (i.e., cisplatin, carboplatin) or pemetrexed according to the respective local labels.
11. Is unable or unwilling to take dexamethasone, folic acid, and/or vitamin B12 supplementation during treatment with pemetrexed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) as Assessed by the Investigator | Up to 5 years

SECONDARY OUTCOMES:
Disease-free Survival Rate | At 2, 3 and 5 years
Overall Survival (OS) | Up to 5 years
Overall Survival Rate | At 2, 3 and 5 years
DFS of Central Nervous System (cDFS) | Up to 5 years
Number of Participants With Treatment Emergent Adverse Events (TEAEs) Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) | Up to 5 years
Number of Participants with Clinically Significant Changes in Clinical Laboratory Parameters | Up to 5 years
Number of Participants with Clinically Significant Changes in Vital Signs | Up to 5 years
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Parameters | Up to 5 years
Number of Participants With Change in Left Ventricular Ejection Fraction (LVEF) Evaluated Using Electrocardiography (ECHO) and Multigated Acquisition (MUGA) Scan | Up to 5 years
Change in EuroQuality of Life-5 Dimensional 3-Level (EQ-5D-3L) | Baseline, up to 5 years
  EQ-5D-3L is a standardized measure of the participant's health-related quality of life (QoL). EQ-5D is a 5-item questionnaire that assesses 5 domains including 1. mobility, 2. self-care, 3. usual activities, 4. pain/discomfort and 5. anxiety/depression. Each dimension has 3 levels ranging from no problems to extreme problems. Higher scores indicate improvement in status of health. The responses will be used to derive overall score using a visual analog scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change From Baseline in European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire-Core 30 (EORTC-QLQ-C30) Scores | Up to 5 years
  EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the global health status/quality of life scale indicates a better level of functioning, and positive changes from baseline indicate improvement.

CONTACTS AND LOCATIONS:
Locations (213):
- United States (13):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - D&H Cancer Research Center - Margate, Margate, Florida
  - Alpha Oncology Research, Orange City, Florida
  - University of Illinois Medical Center, Chicago, Illinois
  - Profound Research LLC at Michigan Hematology and Oncology Consultants, Dearborn, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Perlmutter Cancer Center - 34th Street, New York, New York
  - Memorial Sloan Kettering Cancer Center - New York, New York, New York
  - Atrium Health Wake Forest Baptist - Comprehensive Cancer Center, Charlotte, North Carolina
  - Gabrail Cancer and Research Center, Canton, Ohio
  - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
- Argentina (4):
  - Instituto Argentino de Diagnóstico y Tratamiento, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Centro de Investigación Pergamino SA, Pergamino, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - CEMAIC - Centro de Especialidades Médicas Ambulatorias e Investigación Clínica, Córdoba
- Australia (3):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - GenesisCare - North Shore, St Leonards, New South Wales
  - Saint John of God - Subiaco Hospital, Subiaco, Western Australia
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - Universitair Ziekenhuis (UZ) Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant
- Brazil (25):
  - NOHC - Núcleo de Oncologia e Hematologia do Ceará - José Lourenço, Fortaleza, Ceará
  - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Centro de Pesquisas Clínicas Em Oncologia - CPCO, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Santa Rita, Vitória, Espírito Santo
  - Núcleo de Oncologia da Bahia Ondina - NOB, Salvador, Estado de Bahia
  - Oncoclinicas Oncovida - Brasilia, Brasília, Federal District
  - Cetus Oncologia - Unidade Belo Horizonte, Belo Horizonte, Minas Gerais
  - Cenantron Centro Avançado de Tratamento Oncológico, Belo Horizonte, Minas Gerais
  - Centro Integrado de Oncologia de Curitiba (CIONC), Curitiba, Paraná
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco
  - Centro de Pesquisa Vencer e Oncoclínica - Teresina, Teresina, Piauí
  - Instituto D'Or de Pesquisa e Ensino - Rio de Janeiro, Botafogo, Rio de Janeiro
  - Liga Contra o Câncer - Centro Avançado de Oncologia, Natal, Rio Grande do Norte
  - Clínica Viver, Centro Santa Maria, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia Hospital - Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus - Centro Integrado de Oncologia, Porto Alegre, Rio Grande do Sul
  - Grupo ELORA, Florianópolis, Santa Catarina
  - CHO Centro - Centro de Hematologia e Oncologia de Joinville, Joinville, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos - Hospital de Amor, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto de Oncologia de Sorocaba, Sorocaba, São Paulo
  - A Beneficência Portuguesa de São Paulo, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual, São Paulo
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - William Osler Health System - Brampton Civic Hospital, Montreal, Quebec
- France (22):
  - Hôpital Saint-André, Bordeaux, Aquitane
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - L'Hôpital Nord-Ouest (HNO) - Villefranche-sur-Saône, Villefranche-de-Rouergue, Aveyron
  - Hôpital Côte De Nacre, Caen, Basse-Normandie
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - Hôpital Emile Muller, Mulhouse, Grand Est
  - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire De Nantes - Hôpital Nord Laennec, Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier Universitaire d'Angers, Angers, Maine-et-Loire
  - CHU d Angers, Angers, Maine-et-Loire
  - Institut de Cancérologie de l'Ouest - Angers, Angers, Maine-et-Loire
  - CHU de Nimes - Caremeau Nord, Nîmes, Occitanie
  - Centre Hospitalier Le Mans, Le Mans, Pays de la Loire Region
  - Hopital Prive du Confluet, Nantes, Pays de la Loire Region
  - Hôpital Privé du Confluent, Nantes, Pays de la Loire Region
  - Hopital Nord Ouest, Gleizé, Rhône
  - Gustave Roussy, Villejuif
  - Hôpital Ambroise-Paré, Boulogne-Billancourt, Île-de-France Region
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Île-de-France Region
  - Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region
  - Hôpital Bichat - Claude-Bernard, Paris, Île-de-France Region
- Germany (4):
  - SLK-Kliniken - Fachklinik Löwenstein, Löwenstein, Baden-Wurttemberg
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - Universitätsklinikum Gießen und Marburg - Gießen, Giessen, Hesse
  - Kliniken der Stadt Köln, Cologne, North Rhine-Westphalia
- Greece (5):
  - Saint Savvas Anticancer - Oncological Hospital of Athens, Athens, Attica
  - General Hospital for Thoracic Diseases Sotiria, Athens, Attica
  - Metaxa Cancer Hospital of Piraeus, Athens, Attica
  - BioClinic Thessaloniki, Athens, Central Macedonia
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki, Central Macedonia
- Hong Kong (3):
  - Humanity & Health Clinical Trial Centre, Hong Kong
  - Queen Mary Hospital - Hong Kong, Hong Kong
  - Princess Margaret Hospital, Kowloon
- Italy (24):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola, Forlì-Cesena
  - Azienda Socio Sanitaria Territoriale (ASST) di Bergamo Ovest, Legnano, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan, Milan
  - Istituto Europeo di Oncologia, Milan, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan, Milan
  - Ospedale del Mare, Napoli, Naples
  - Ospedale Santa Maria delle Croci di Ravenna, Lugo, Ravenna
  - Azienda Ospedaliera Complesso Ospedaliero San Giovanni - Addolorata, Roma, Rome
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Ospedale P. Pederzoli - Casa di Cura Privata S.p.A., Peschiera del Garda, Verona
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo - Alessandria, Alessandria
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Humanitas Gavazzeni, Bergamo
  - Azienda Socio Sanitaria Territoriale (ASST) Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico Sant Orsola-Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Policlinico Gaspare Rodolico - San Marco - Catania/ Presidio G. Rodolico, Catania
  - Azienda Unita Sanitaria Locale toscana Nord Ovest, Livorno
  - Azienda Unità Sanitaria Locale Toscana Nord Ovest, Livorno
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero - Universitaria di Modena, Modena
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Senese - L'ospedale Santa Maria alle Scotte, Siena
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (17):
  - Aichi Cancer Center, Nagoya, Aiti [Aichi]
  - Kurume University Hospital, Kurume-Shi, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hirosima [Hiroshima]
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Hukuoka [Fukuoka]
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Osakasayama-Shi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Sizuoka [Shizuoka]
  - National Cancer Center Hospital East, Kashiwa-shi, Tiba [Chiba]
  - Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka
- Malaysia (5):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Pulau Pinang, Pulau Pinang, Pulau Pinang
  - Hospital Picaso, Petaling Jaya, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Sunway Medical Centre, Selangor Darul Ehsan
- Mexico (3):
  - Preparaciones Oncológicas S.C., León, Guanajuato
  - Centro Oncológico Alianza XXI, Mexico City, Mexico City
  - Clínica Integral Internacional de Oncología S de RL de CV, Mirador, Puebla
- Netherlands (3):
  - Ziekenhuis St Jansdal Harderwijk, Harderwijk, Gelderland
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Leids Universitair Medisch Centrum (LUMC), Leiden, South Holland
- Peru (3):
  - Hospital Nacional Arzobispo Loayza, Lima Cercado, Lima region
  - IPOR - Instituto Peruano de Oncología & Radioterapia - Sede Principal, San Isidro, Lima region
  - Detecta Clínica, Surquillo, Lima region
- Poland (5):
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin, Greater Poland Voivodeship
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ, Wroclaw, Lower Silesian Voivodeship
  - Mruk-Med I Sp. z o.o., Rzeszów, Podkarpackie Voivodeship
  - Warmińsko-mazurskie Centrum Chorób Płuc w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - Wojewódzki Szpital Specjalistyczny w Białej Podlaskiej, Biała Podlaska
- Romania (7):
  - Institutul Oncologic Bucuresti - Prof. Dr. Alexandru Trestioreanu, Bucharest, Bucharest
  - Monza Oncology Day Hospital, Bucharest, București
  - Centrul de Radioterapie Amethyst Cluj, Floreşti, Cluj
  - Ovidius Clinical Hospital, Ovidiu, Constanța County
  - Clinica MC Gral Ploiesti, Ploieşti, Prahova
  - Oncocenter - Oncologie Clinica, Timișoara, Timiș County
  - Spitalul Județean de Urgență Satu Mare, Satu Mare
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore, North East
  - National Cancer Centre Singapore, Singapore
- South Korea (21):
  - Kyungpook National University Chilgok Hospital, Daegu, Daegu Gwang'yeogsi [Taegu-Kwangyokshi]
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Catholic University of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, Gyeonggido [Kyonggi-do]
  - National Cancer Center - Korea, Goyang-si, Gyeonggido [Kyonggi-do]
  - Keimyung University Dongsan Hospital, Daegu, Gyeongsangbugdo [Kyongsangbuk-do]
  - Kosin University Gospel Hospital, Pusan, Gyeongsangnam-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnamdo [Kyongsangnam-do]
  - Inha University Hospital, Incheon, Incheon Gwang'yeogsi [Inch'on-Kwangyokshi]
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Jeonbuk National University Hospital, Jeonju, Jeonrabugdo [Chollabuk-do]
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Severance Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Konkuk University Medical Center, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Hanyang University Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
- Spain (15):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Català d'Oncologia Badalona, Badalona, Barcelona
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Instituto Oncológico Dr Rosell, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitario Clínico San Cecilio PTS, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quirónsalud Málaga, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- Thailand (5):
  - Chulabhorn Hospital, Bang Kapi, Bangkok
  - Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok
  - Lampang Cancer Hospital, Muang, Changwat Lampang
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - Navamindradhiraj University - Faculty of Medicine Vajira Hospital, Bangkok, Khet Dusit
- Turkey (Türkiye) (17):
  - Başkent Üniversitesi Adana Dr Turgut Noyan Uygulama ve Araştirma Merkezi, Yüreğir, Adana
  - Ankara Il Saglik Mudurlugu SBU Gulhane Egitim Ve Arastirma Hastanesi, Etlik, Ankara
  - Dicle Üniversitesi Tıp Fakültesi, Sur, Diyarbakır
  - Gaziantep Universitesi - Şahinbey Araştırma ve Uygulama Hastanesi, Şehitkamil, Gaziantep
  - Memorial Bahçelievler Hospital, Bahçelievler, Istanbul
  - İstinye Üniversite Hastanesi Liv Hospital Bahcesehir, Esenyurt, Istanbul
  - İ.A.Ü. VM Medical Park Florya Hastanesi, Küçükçekmece, Istanbul
  - Medicana International Izmir Hastanesi, Turgutlu, Manisa
  - VM Medical Park Samsun Hastanesi, Atakum, Samsun
  - Medical Park Seyhan Hastanesi, Adana
  - T.C. Saglik Bakanligi Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Liv Hospital Ankara, Ankara
  - Trakya Üniversitesi Sağlık Araştırma ve Uygulama Merkezi, Edirne
  - Ozel Gaziantep Medical Point Hastanesi, Gaziantep
  - T.C. Saglik Bakanligi - Istanbul Il Saglik Mudurlugu - Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
- United Kingdom (3):
  - The Christie NHS Foundation Trust, Manchester, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Velindre University NHS Trust, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: No